CLINICAL TRIAL: NCT04007731
Title: Effects of New Protein Bar on Biochemical and Physiological Parameters in Physically Active People
Brief Title: New Protein Bar for Physically Active People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zala Jenko Praznikar (Other)
Responsible Party: Sponsor-Investigator, Zala Jenko Praznikar, assistant professor, University of Primorska
Organization: University of Primorska (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: barsport
Record Dates: First submitted 2019-06-21; First posted 2019-07-05 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Muscle Mass; Inflammation; Regeneration Muscle
Keywords: protein bar; physical activity; muscle
MeSH Terms: conditions — Inflammation; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein, high fibre and creatine load bar (DrRip) (Experimental): 1 new protein bar (260 kcal) after training every day
  Interventions: Dietary Supplement: DrRip - high protein, high fibre and creatine load
- Voltage energy bar (Active Comparator): 1 control commercially available protein bar (260 kcal) after training every day
  Interventions: Dietary Supplement: Voltage energy bar

INTERVENTIONS:
Dietary Supplement: DrRip - high protein, high fibre and creatine load — A protein bar or control bar consumption after training every day for 5 days, 5 days wash-out, 5 days second bar consumption
  Other Names: Protein product
  Arms: High protein, high fibre and creatine load bar (DrRip)
Dietary Supplement: Voltage energy bar — A protein bar or control bar consumption after training every day for 5 days, 5 days wash-out, 5 days second bar consumption
  Other Names: control protein bar
  Arms: Voltage energy bar

SUMMARY:
Post-exercise nutrition is an important factor in a nutrition plan for physically active subjects. Focusing on that, the Serbian group is developing protein bars enriched with sports supplements. Slovenian partner group will investigate the effect of new protein bar consumption on body composition, biochemical parameters, and muscle regeneration after training. The new bar will be compared with a commercially available bar.

DETAILED DESCRIPTION:
The clinical study will be performed on 10 elite handball players from Slovenia handball club. It will be designed as a crossover study. Half of the participants will consume the new bar for five days and the other half will consume the control bar. After the five-day washout period, the groups will consume the bar which was not consumed in the first period.

At baseline, at the end of every intervention and washout period, the blood samples will be withdrawn, and the body composition will be analyzed.

The analyzed biochemical parameters will be basic serum parameters, such as fasting glucose, total cholesterol, LDL, HDL, triglycerides, aspartate aminotransferase (AST), alanine aminotransferase (ALT), C-reactive protein (CRP), and parameters related to the muscle regeneration and inflammation, such as creatine kinase, lactate dehydrogenase, insulin-like growth factor (IGF), tumor necrosis factor alpha (TNF-alpha), interleukin 6 (IL-6), monocyte chemoattractant protein 1 (MCP-1).

In the second part of the study, the acute effect of consuming each bar after training will be tested. Each participant will consume both bars on separate days. The mentioned parameters will be assessed after training and immediately and 3h after bar consumption.

ELIGIBILITY:
Inclusion Criteria:

* daily high-intensity physical activity

Exclusion Criteria:

* smoking, cardiovascular, neurological, skeletal muscle disease, allergies

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 10 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Muscle mass | 15 days
  Muscle mass in kilograms will be determined using bioelectrical impedance analysis (BIA).
Fat mass | 15 days
  Fat mass in kilograms will be determined using bioelectrical impedance analysis (BIA).

SECONDARY OUTCOMES:
C-reactive protein | 15 days
  Serum levels of C-reactive protein (parameter of inflammation) will be analyzed by biochemistry analyzer (Cobass c111).
Creatine kinase | 15 days
  Serum levels of creatine kinase (marker of regeneration) will be analyzed by biochemistry analyzer (Cobass c111).
Lactate dehydrogenase | 15 days
  Serum levels of creatine kinase (marker of regeneration) will be analyzed by biochemistry analyzer (Cobass c111).
Tumor necrosis factor alpha | 15 days
  Serum levels of Tumor necrosis factor alpha (parameter of inflammation) will be analyzed by enzyme linked immunosorbent assays (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No
Other researchers on the study (Saša Kenig, Ana Petelin, Tadeja Jakus) will analyze samples, which will be coded by PI